CLINICAL TRIAL: NCT01455688
Title: Early Antiretroviral Therapy for Critically Ill HIV Infected Patients
Brief Title: Early Antiviral Therapy for Critically Ill HIV Infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Marcio Manozzo Boniatti, Principal investigator, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARV-0112
Record Dates: First submitted 2011-10-17; First posted 2011-10-20 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: HIV Infection
Keywords: critically ill patients; HIV infection; HAART; mortality
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early antiviral therapy (Experimental)
  Interventions: Drug: early HAART
- Conventional therapy (Active Comparator)
  Interventions: Drug: Late HAART

INTERVENTIONS:
Drug: early HAART — Initiation of HAART within 5 days of ICU admission
  Arms: Early antiviral therapy
Drug: Late HAART — Initiation of HAART after ICU discharge
  Arms: Conventional therapy

SUMMARY:
The aim of the study is to verify the effect of HAART in critically ill HIV infected patients. The current practice is to begin antiviral therapy after ICU discharge, when the condition of the patient is more stable. The investigators hypothesis is that the investigators can improve outcome of these patients with earlier antiviral therapy in the ICU. The investigators just have retrospective studies in this scenario. After admission to ICU, patients are assigned to one of two arms: early HAART (within 5 days of ICU admission) or conventional therapy (initiation of HAART after ICU discharge). The following data will be collected: demographic variables, CD4 count, viral load, drug toxicity, opportunistic infection, hemodialysis, mechanical ventilation and vasoactive drug. The patients will be followed to determine ICU mortality, hospital mortality and 6-month mortality.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* CD4 cell count less than 350 cells/mm3 within 3 months prior to study entry OR CD4 cell count between 350 cells/mm3 and 500 cells/mm3 if age > 55 years, coinfection with HBV or HCV, neoplasia, viral load > 100,000 copies/ml or elevated cardiovascular risk OR AIDS-defining illness

Exclusion Criteria:

* Regular use of HAART
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Hospital mortality | 4 weeks
  It is a estimative of length of hospital stay

SECONDARY OUTCOMES:
6-month mortality | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Boniatti MM, Pellegrini JAS, Marques LS, John JF, Marin LG, Maito LRDM, Lisboa TC, Damiani LP, Falci DR. Early antiretroviral therapy for HIV-infected patients admitted to an intensive care unit (EARTH-ICU): A randomized clinical trial. PLoS One. 2020 Sep 21;15(9):e0239452. doi: 10.1371/journal.pone.0239452. eCollection 2020. PMID 32956419